CLINICAL TRIAL: NCT06954857
Title: The Influence of Standardized Process Management of Laryngeal Mask Airway Placement Based on Pressure Monitoring on the Incidence of Adverse Reactions in Elderly Patients During the Perioperative Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanqi Yang (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor-Investigator, Xuanqi Yang, Resident physicians, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-218-01
Record Dates: First submitted 2025-04-03; First posted 2025-05-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: LMA; Pressure Injury; Elderly; Airway Management
Keywords: Laryngeal Mask Airway (LMA); Pressure Monitoring; Elderly Patients; Complications; ERAS
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: the pressure was monitored and adjusted in real time (Experimental): The measured and adjusted airway pressure, cuff pressure and leak pressure were recorded
  Interventions: Device: Cuff pressure monitor
- Control group：the pressure was measured once after empirical inflation of the laryngeal mask (No Intervention): The cuff pressure, airway pressure, and leak pressure were measured only once after empirical inflation under the condition of guaranteed ventilation

INTERVENTIONS:
Device: Cuff pressure monitor — Participants were allocated to the experimental group and the control group using block randomization.
  Experimental group: A pressure monitor was used to continuously monitor and promptly adjust the cuff pressure, seal pressure, and leakage pressure of the laryngeal mask.
  Arms: Experimental group: the pressure was monitored and adjusted in real time

SUMMARY:
The laryngeal mask airway (LMA) is a supraglottic ventilation device designed according to human anatomy. It was developed in 1981 by Dr. Archie Boubrain in the United Kingdom to compensate for the deficiencies of tracheal intubation and mask ventilation. It has been widely used in clinical practice because of its simple operation, small airway stimulation, and hemodynamic stability. In 1990, LMA entered the Chinese market. In 1993, LMA was included in the American Society of Anesthesiologists guidelines for the emergency management of the difficult airway. In the past, tracheal intubation was the standard method of airway control during general anesthesia. In the past decade, the proportion of LMA ventilated general anesthesia has increased significantly in China and European and American countries. By 2022, the utilization rate of LMA in China climbed to 95.96%. With the continuous improvement and development of LMA, it can be used to establish safe airway management in special positions such as lateral position and prone position, long-term surgery and special site surgery.

However, the wide application has also exposed some key problems. The lack of standardized process management of LMA placement may lead to improper placement, airway obstruction, laryngspasm, reflux, and aspiration during the application of LMA, which may cause a series of pulmonary and extrapulmonary complications. Studies have shown that many adverse events during LMA implantation may be related to LMA pressure monitoring. Inadequate pressure monitoring may lead to pressure imbalance, and improper pressure management may lead to poor coordination between LMA and pharynx. Coupled with the change in intraoperative position and postoperative transfer, the risk of postoperative sore throat and LMA displacement increases. Therefore, there is an urgent need for standardized process management, dynamic pressure monitoring and position adjustment during the use of LMA. The standardized management of LMA insertion involves the standardized selection, placement, maintenance management and transportation of LMA. Especially for the elderly population, LMA displacement is more likely to occur due to the atrophy of pharyngeal mucosa and muscle, weakened cough reflex, and decreased chest wall compliance, which increases the incidence of pulmonary and extrapulmonary complications. For elderly patients with atherosclerosis, LMA displacement and relatively high cuff pressure may compress the jugular and jugular veins in the neck and surrounding tissues, increasing the risk of stroke in elderly patients. Effective and safe anesthesia airway and respiratory management strategies during general anesthesia will directly affect the occurrence of postoperative pulmonary complications (PPCs) and the incidence of sore throat in elderly patients. Standardized management of LMA and continuous pressure monitoring and adjustment can improve the above adverse reactions.

At present, there is a lack of large-scale and reliable evidence-based medical evidence to evaluate the effect of standardized process management of laryngeal mask insertion based on pressure monitoring on perioperative adverse reactions in elderly patients with high risk of pulmonary complications. Especially in the elderly population with a high incidence of PPCs, the safety, short - and long-term advantages and disadvantages of widespread use of LMA ventilation are still unclear. Therefore, it is particularly urgent to carry out the effect of standardized process management of laryngeal mask insertion based on pressure monitoring on perioperative adverse reactions in elderly patients, and to further explore the appropriate range of laryngeal mask related pressure indicators. This study based on the concept of enhanced recovery after surgery (ERAS) can not only fill the current research gap, but also provide strong support for safe and efficient airway management in elderly patients during the perioperative period, and effectively promote the further optimization of clinical practice, which has extremely important clinical significance and practical value.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) is a supraglottic ventilation device designed based on human anatomy. It was developed by Dr. Archie Brain from the UK in 1981 to compensate for the deficiencies of tracheal intubation and mask ventilation . Due to its advantages such as simple operation, minimal irritation to the airway, and more stable hemodynamics, it has been widely used clinically. In 1990, the LMA entered the Chinese market. In 1993, it was included in the ASA Guidelines for the Management of the Difficult Airway. In the past, endotracheal intubation was the standard method for airway control during general anesthesia. The proportion of general anesthesia using LMA ventilation has also increased significantly in China, Europe, and the United States in the past decade. By 2022, the popularization rate of LMA use in China had climbed to 95.96%. With the continuous improvement and development of the LMA, a safe airway can be established through the LMA in special positions such as the lateral or prone position, as well as in long - term and special - site surgeries. Goldmann et al. conducted animal experiments and concluded that it is feasible to keep the LMA inserted for up to 8 hours when the LMA pressure is appropriate. It can be seen that the LMA has become a widely used airway management tool in clinical medicine.

However, wide application has also exposed key problems. The lack of standardized process management for LMA placement may lead to improper placement, airway obstruction, laryngospasm, regurgitation, and aspiration during its application, resulting in a series of pulmonary and extrapulmonary complications. Studies have shown that many adverse events during LMA placement may be related to LMA pressure monitoring. The lack of pressure monitoring can lead to pressure imbalance . Unreasonable pressure management may cause poor fitting between the LMA and the pharynx. Coupled with changes in body position during surgery and postoperative transfer, the risks of postoperative sore throat and LMA displacement increase. Therefore, there is an urgent need for dynamic pressure management and body - position adaptability adjustment during LMA use.

First, in the pressure management of the LMA, the precise control of cuff pressure is the core. Cuff pressure is defined as the pressure inside the cuff of the LMA ventilation mask after gas is filled, which is related to factors such as cuff inflation volume, LMA model, and temperature. For inflatable LMAs, clinically, a syringe is often used empirically to inflate the inflation balloon and valve on the LMA one - way valve. The inflation status of the ventilation mask cuff is judged by the inflation status of the balloon on the one - way valve. It is considered appropriate when the LMA does not leak air, and the tidal volume and peak airway pressure are within the normal range. Too low cuff pressure may lead to poor ventilation, while too high pressure can compress the pharyngeal mucosal tissue, resulting in postoperative pharyngeal complications. In addition, the inhalation of N₂O during clinical anesthesia can increase the cuff pressure. Therefore, regular monitoring of cuff pressure is of great significance . Previous clinical studies have used self - made cuff pressure gauges to monitor LMA cuff pressure and set the LMA cuff pressure based on the peak airway pressure. These studies have shown that appropriate inflation volume under cuff pressure monitoring and setting the cuff pressure at Ppeak + 0 - 5cmH₂O during general anesthesia with LMA ventilation can produce a good sealing effect and reduce the incidence of postoperative pharyngeal complications. Research on the reasonable inflation volume of the LMA cuff shows that low - pressure cuff inflation of the LMA is beneficial for the rapid postoperative recovery of patients .

Secondly, the sealing pressure and leakage pressure of LMA are greatly affected by the head and neck. Therefore, adaptive adjustment of position is of great significance for laryngeal mask pressure management. The sealing pressure is the pressure required to create an effective seal between the LMA and the surrounding laryngeal tissue. It is formed by the matching and extrusion of laryngeal mask and periglottic pharyngeal tissue structure, which can reflect the alignment of laryngeal mask and the degree of fitting to the pharynx, and is related to the type of laryngeal mask and the laryngeal structure of the patient. The current LMA is divided into three generations according to whether it has esophageal drainage and visual function. The first-generation LMA was a single-tube LMA with a sealing pressure less than 20cmH₂O. On the basis of the first generation, the second generation LMA added an esophageal drainage tube, and the sealing pressure was up to 30cmH₂O. On the basis of the second generation, the third generation LMA added a video endoscope channel, and the sealing pressure was 25-30 CMH ₂O. Appropriate LMA sealing pressure can ensure airway sealing and maintain normal respiratory function. The leakage pressure is the pressure at which gas leaks from the edge of the LMA as the airway pressure gradually rises. The oropharyngeal leakage pressure is often used clinically to assess the reliability of the LMA seal during actual ventilation. Studies have shown that oropharyngeal leak pressure is the most accurate description of the gas leak pressure around the oropharynx, which is related to many factors such as the anatomical structure of the patient's upper airway, anesthetic drugs, laryngeal mask model, and surgical position. The higher the oropharyngeal leakage pressure, the better the alignment and fit of the LMA to the pharynx. Air leakage around the laryngeal mask can lead to hypoventilation and even increase the risk of reflux and aspiration. Studies have shown that a variety of factors such as pharyngeal anatomy, head and neck position, and surgical position can cause LMA displacement and affect ventilation. Moderate flexion of the head and neck can increase the oropharyngeal leak pressure, while extension or rotation can reduce the oropharyngeal leak pressure. The neutral position is between the two. Excessive flexion may lead to a significant increase in airway pressure or airway obstruction, affecting ventilation. The use of 45° head position rotation during laparoscopic surgery in children does not affect effective ventilation, and can reduce leakage pressure and laryngeal mask displacement. Some studies have also proposed that the head swing amplitude should be less than 10 to 15° when moving the head during surgery. Chandan et al. found that the laryngeal mask cuff was optimally positioned after LMA insertion in 56.7% of patients, but non-optimally positioned did not affect normal and effective ventilation. A few severe cases can cause hypoxemia and carbon dioxide retention. The shear force generated during postoperative transfer of laryngeal mask is also an independent risk factor for laryngeal mask displacement caused by postural change. The combined effect of postural change and metastasis may cause laryngeal mask microdisplacement, resulting in delayed ventilatory impairment. New research devices have been developed to prevent LMA displacement affecting ventilation during transfer.

Therefore, standardized process management for LMA placement and ensuring reasonable LMA pressure to maintain correct LMA alignment and effective ventilation function are extremely important. However, currently, clinical practice does not mandate the monitoring of LMA pressure indicators such as cuff pressure. There is no unified standard for pressure measurement, limited research on LMA pressure values in different body positions, and the optimal values of various LMA pressures are not clear. Previous studies have explored the reasonable inflation volume of the LMA cuff, defining the optimal cuff inflation volume as the volume that meets the requirements of positive - pressure ventilation greater than 17cmH₂O, an LMA cuff pressure of 40 - 80cmH₂O, and an oropharyngeal leakage pressure greater than 20cmH₂O. However, these studies were limited to size 4 LMAs. Regarding the use of pressure gauges to monitor cuff pressure, a study compared the accuracy of the hand - touch method, passive release method, and minimum occluding volume method in tracheal tube cuff pressure monitoring, indicating that the passive release method has the highest accuracy in cuff pressure control. In this regard, Wang et al. developed a mobile terminal application that can monitor and adjust tracheal tube cuff pressure in real - time, which can maintain the cuff pressure within a reasonable range and significantly reduce the incidence of postoperative adverse reactions. Whether such methods are applicable to LMA pressure monitoring remains to be further explored. The expert consensus on the clinical application and management of the LMA also indicates the importance of measuring LMA - related pressures such as cuff pressure, sealing pressure, and leakage pressure.

Especially for the elderly population, due to the atrophy of pharyngeal mucosa, weakened cough reflex, and decreased chest wall compliance, they are at high risk of postoperative pulmonary complications. Effective and safe anesthetic airway and respiratory management strategies during general anesthesia will directly affect the occurrence of postoperative pulmonary complications (PPCs) and the incidence of sore throat in the elderly. Our research group has previously completed the design and production of an air - cuff pressure monitoring device. The investigators speculate that the application of standardized process management for LMA placement under pressure monitoring in elderly patients at high risk of postoperative pulmonary complications can reduce the incidence of LMA displacement, postoperative sore throat, and PPCs. Currently, there is a lack of large - scale and reliable evidence - based medical evidence to evaluate the impact of standardized process management for LMA placement based on pressure monitoring on perioperative adverse reactions in elderly patients at high risk of pulmonary complications. Especially, the safety and short - and long - term benefits and drawbacks of extensive use of LMA ventilation in the elderly population with a high incidence of PPCs are unclear. Therefore, it is necessary to conduct a prospective, randomized controlled study to explore the impact of standardized process management for LMA placement based on pressure monitoring compared with conventional inflatable LMAs on LMA displacement, sore throat, and pulmonary complications in elderly patients during the perioperative period. Combined with dynamic monitoring, the risk of LMA displacement can be noticed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years old
* Non-cardiothoracic surgery and head and neck surgery
* Elective surgery
* ASA I-III grade
* NYHA cardiac function class I-II
* The operation time is expected to be ≥30 minutes and ≤2 hours
* 18.5≤BMI (kg/m2) ≤24.9

Exclusion Criteria:

* Change to emergency surgery
* Difficult airway that can be predicted before operation, such as difficulty in opening mouth and limited neck movement
* Loose teeth
* Laryngeal obstruction, laryngeal edema, laryngeal abscess, acute airway inflammation, full stomach, acute abdomen, abdominal trauma, drug poisoning, gastrointestinal bleeding
* Complicated with chronic obstructive pulmonary disease, asthma and other respiratory diseases
* Allergic to laryngeal mask materials
* Non-supine position
* Inability to cooperate with the investigator for any reason
* Taking other investigational drugs or participating in other clinical trials within 3 months before study entry
* The investigators considered it inappropriate to be included in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of sore throat | 10 minutes, 1 hour, 2 hours, 24 hours, and 48 hours after LMA removal
  VAS scale was used to evaluate the scores. The scale consisted of a 10-cm straight line, with the left end of the line indicating "no pain" and the right end indicating "severe pain". A total of 6 different degrees of facial expressions were used to express the degree of pain, including no pain, slight pain, mild pain, moderate pain, severe pain and severe pain.
  In this study, sore throat was considered to occur as long as VAS≥3 points at any evaluation time point after LMA removal.

SECONDARY OUTCOMES:
The incidence of intraoperative laryngeal mask displacement | intraoperatively
  In this study, LMA displacement was considered as long as "glottis not seen" or "the epiglottis touched the glottic fissure and the glottis was visible" was observed under fiberoptic bronchoscopy。
The incidence of pulmonary complications within 7 days after surgery | within 7 days after surgery
  According to the symptoms and corresponding diagnostic criteria. Hypoxemia is defined as: Arterial PaO2 < 60mmHg or SpO2 < 90%, in which mild hypoxemia was arterial PaO2 60-79 MMHG or SpO2 90%-94%, moderate hypoxemia was arterial PaO2 40-59 MMHG or SpO2 85%-89%, and mild hypoxemia was arterial PaO2 60-79 MMHG or spo2 90%-94%. Severe hypoxemia was defined as arterial PaO2 < 40mmHg or SpO2 < 85%. Carbon dioxide retention was defined as arterial PaCO2 greater than 45mmHg, with mild carbon dioxide retention: 45 to 50mmHg, moderate carbon dioxide retention: 50 to 70mmHg, and severe carbon dioxide retention: PaCO2 > 70mmHg. Atelectasis was diagnosed by bedside chest radiography or CT. The diagnosis of pneumonia was based on the standard of the Centers for Disease Control and Prevention of the United States. The diagnosis of ARDS was based on the Berlin definition criteria.
The length of hospital stay | within 7 days after surgery
  The length of hospital stay by consulting the hospitalization system
The score of Laryngeal mask alignment | Within 5 minutes after laryngeal mask placement
  Keller's grading system, a method used to assess the alignment of the laryngeal mask, scores the glottis and epiglottis by looking at how visible they are, as follows:
  Grade 1: Glottis not seen, which indicates poor alignment of the LMA and may require further adjustment.
  Grade 2: The epiglottis touched the glottic fissure and the glottis was visible, indicating that the position of the LMA had improved somewhat but was still not optimal.
  Grade 3: Both epiglottis and glottis are visible, at which point the LMA is in good alignment.
  Grade 4: only glottis is seen, which is the best position, indicating that the LMA is in an ideal position and can provide good airway support for the patient.
Arterial partial pressure of oxygen | perioperative period
The changes of inflammatory factors | Before surgery and on the first day after surgery
  Venous blood was collected for blood routine test, and the changes of inflammatory factors were recorded
The total cost by consulting the hospitalization system | within 7 days after surgery
Arterial partial pressure of carbon dioxide | perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No